CLINICAL TRIAL: NCT05386238
Title: Engaging Men From Blue-collar Industries in Weight Loss: Study 3- Evaluating the Acceptability of Weight Loss Treatments
Brief Title: Engaging Men From Blue-collar Industries in Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Melissa M. Crane, PhD, Assistant Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18013105-IRB01
Record Dates: First submitted 2022-05-12; First posted 2022-05-23 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Obesity
Keywords: occupation; Behavioral treatment
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored treatment (Experimental): 6-months of group-based behavioral weight loss treatment tailored to men working in blue-collar occupations.
  Interventions: Behavioral: Tailored behavioral weight loss program
- Standard of care treatment (Active Comparator): 6-months of group-based behavioral weight loss treatment following the Diabetes Prevention Program Group Lifestyle balance.
  Interventions: Behavioral: Standard behavioral weight loss program

INTERVENTIONS:
Behavioral: Standard behavioral weight loss program — 16 internet-delivered, group sessions over 6 months supported by digital handouts. The intervention will focus on changes to eating, physical activity, and self-monitoring.
  Arms: Standard of care treatment
Behavioral: Tailored behavioral weight loss program — 16 internet-delivered, group sessions over 6 months supported by digital handouts or videos tailored to men working in blue-collar occupations. The intervention will focus on changes to eating, physical activity, and self-monitoring.
  Arms: Tailored treatment

SUMMARY:
Objectives*: Primary Objective: Aim 1: Examine the acceptability of tailored behavioral weight loss program and a standard program in men working in blue-collar occupations.

Aim 2: Compare recruitment approaches that vary on trust-based messaging to recruit men with overweight/obesity who work in blue-collar occupations.

Secondary Objectives: Determine the feasibility of retaining participants to a randomized trial over six months.

DETAILED DESCRIPTION:
Men working in blue-collar occupations have a high prevalence of overweight and obesity and have high rates of comorbidities associated with obesity. Unfortunately, these men are unlikely to participate in evidenced-based weight loss interventions. Further, few efficacious interventions have been developed that target this population for weight control. The purpose of this study is to test the feasibility and acceptability of tailored recruitment messages and a novel, tailored behavioral weight loss intervention in the context of a randomized trial.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 years and older
2. Male
3. Body mass index (BMI) > 25 kg/m2
4. Employed >20 hours per week in an occupation classified as blue collar
5. Ability to communicate in English
6. Provision of signed and dated informed consent form

Exclusion criteria:

1. History of bariatric surgery
2. Diabetes managed with insulin
3. Diagnosis of a serious mental illness
4. Conditions contraindicated to exercise independently (determined using four questions of Physical Activity Readiness Questionnaire)
5. Report of potentially hazardous alcohol use (ASSIST >27)
6. Weight loss in the prior six months of 10 pounds or greater
7. Body mass index ≥60 kg/m2, due to increased injury risk with exercise
8. Diagnosis of an eating disorder
9. Any major medical condition that could increase risk for injury or other contradictions for treatment, or high likelihood of attrition, as determined by the study team

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as male
Enrollment: 28 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa M Crane, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Crane MM, Feit C, Yeh C, Ortiz MG, Appelhans BM. Feasibility and Acceptability of Behavioral Weight Loss Programs for Men in Trade and Labor Occupations: A Pilot Study. Obes Sci Pract. 2025 Mar 1;11(2):e70066. doi: 10.1002/osp4.70066. eCollection 2025 Apr. PMID 40918631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between September 28, 2022, and March 30, 2023. Recruitment was closed before our planned sample size was recruited to complete the study within the funding period
Pre-assignment Details: All consented participants were randomized into the study. 63 who completed the initial screening were excluded due to not meeting eligibility criteria, 9 were unable to be contacted, and 17 did not complete the study enrollment procedures.
Period: Overall Study
Arm/Group | Tailored Treatment | Standard of Care Treatment
Started | 14 | 14
Completed | 11 | 11
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Treatment | Standard of Care Treatment | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44.5 [38 to 53] | 44 [40 to 55] | 44 [38.5 to 54.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 8 | 7 | 15
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 14 | 28
BMI (kg/m2) [Median (Inter-Quartile Range); unit: kg/m2] | 31.6 [31.2 to 43.3] | 33.4 [31.1 to 39.6] | 31.8 [31.1 to 39.6]

OUTCOME MEASURES:

1. Primary Outcome: Participant Satisfaction With the Intervention
Description: Acceptability of the intervention will be reported as participants' satisfaction with the program rated on a 4-point scale. "How satisfied are you overall with the weight management program you received from the Study?"
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Treatment | Standard of Care Treatment
Number analyzed (Participants) | 12 | 11
Participants
  Very Dissatisfied | 2 | 1
  Dissatisfied | 0 | 0
  Somewhat Satisfied | 3 | 2
  Very Satisfied | 7 | 8

2. Primary Outcome: Recruitment Response
Description: The proportion of participants who enroll in the study by recruitment message type.
Time Frame: Baseline
Population: 1000 postcards of each message type were sent to men in the recruitment area. A subset of postcards were returned undelivered and were removed from the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Message: The general recruitment message emphasized improving energy, a common goal for men initiating weight loss that was identified during preparatory work.
- Enhanced Trust: The enhanced trust recruitment message emphasized the formative work conducted prior to the development of the intervention and the standard recruitment message.
- Endorsement: The recruitment message included a quote from a prior participant indicating satisfaction with the program and the standard recruitment message.
- Combined: Combined the standard recruitment message with the enhanced trust and endorsement messages.
Arm/Group | Standard Message | Enhanced Trust | Endorsement | Combined
Number analyzed (Participants) | 906 | 942 | 915 | 931
Participants | 3 | 1 | 3 | 0

3. Secondary Outcome: Retention Rates for Each Intervention Group
Description: Proportion of participants who complete the final follow up assessment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Treatment | Standard of Care Treatment
Number analyzed (Participants) | 14 | 14
Participants | 11 | 11

4. Secondary Outcome: Recruitment Reach
Description: Number of visits to study websites
Time Frame: Baseline
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Message | Enhanced Trust | Endorsement | Combined
Number analyzed (Participants) | 906 | 942 | 915 | 931
Participants | 34 | 14 | 17 | 9

5. Other Pre Specified Outcome: Clinically Significant Weight Loss
Description: Proportion of participants who achieve a weight loss >5% of initial weight
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Treatment | Standard of Care Treatment
Number analyzed (Participants) | 14 | 14
Participants | 4 | 4

6. Other Pre Specified Outcome: Program Perceptions
Description: Semi-structured interviews to evaluate participants perceptions of program
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Collected at 3 and 6 months assessments systematically and as reported by participants during intervention visits
Arm/Group | Tailored Treatment | Standard of Care Treatment
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tailored Treatment (N=14) | Standard of Care Treatment (N=14)
Emergency room visit (General disorders) | 0 | 2
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT05386238/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT05386238/ICF_001.pdf